CLINICAL TRIAL: NCT03322267
Title: A Single-arm Phase II Study of Chemoradiotherapy Plus Pembrolizumab as Adjuvant Therapy for Locally Advanced Esophageal Squamous Cell Carcinoma Patients at High Risk of Recurrence Following Preoperative Chemoradiotherapy Plus Surgery
Brief Title: Adjuvant Pembrolizumab for Patients With Locally Advanced Esophageal Squamous Cell Carcinoma at High Risk of Recurrence
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201708042MIPD
Record Dates: First submitted 2017-10-16; First posted 2017-10-26 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-09

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Adjuvant pembrolizumab; Chemoradiotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — pembrolizumab; Cisplatin; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Adjuvant cisplatin-chemoradiotherapy followed by pembrolizumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab (Experimental): Adjuvant cisplatin-chemoradiotherapy followed by pembrolizumab
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Cisplatin (30 mg/m2, QW, 2 cycles) and radiotherapy (18-26 Gy/10-13 fractions) as adjuvant chemoradiotherapy, followed by pembrolizumab (200mg, Q3W, 18 cycles)
  Other Names: cisplatin; radiotherapy

SUMMARY:
In this study, participants with histologically diagnosed locally advanced esophageal squamous cell carcinoma who have received preoperative cisplatin-based chemoradiotherapy followed by surgery harbouring high risk of tumor recurrence will receive adjuvant cisplatin-based chemoradiotherapy followed by pembrolizumab. The primary study hypothesis is that adjuvant pembrolizumab will improve the 1-year recurrence-free survival rate compared to historical control.

DETAILED DESCRIPTION:
It is a single-arm phase II trial. The target population is patients with histologically diagnosed locally advanced ESCC patients (clinically staged at least T3 and/or any N and M0 by endoscopic ultrasonography [EUS] and fludeoxyglucose-positron emission tomography [FDG-PET]) who have received preoperative cisplatin-based chemoradiotherapy (CRT) followed by surgery, and exhibit high risk (closed or involved resection margin or extranodal invasion of involved lymph nodes or ypN2-3) of tumor recurrence. Eligible patients will receive adjuvant cisplatin-based CRT followed by pembrolizumab for 18 cycles.The study will enroll 46 patients in Taiwan. The estimated enrollment period is 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be ≥ 20 years of age on day of signing informed consent.
3. Be a diagnosed by pathology or cytology with a locally advanced ESCC, which is clinically stage according to the TNM system of the American Joint Committee on Cancer (AJCC) Cancer Staging System (7th edition), fulfilling one of the following criteria as determined by endoscopic ultrasound, computed tomography, bronchoscopy and positron emission tomography:

   1. T3, N0, M0;
   2. T4a, N0, M0;
   3. T1-4a, N1-3, M0.
4. Have been treated with preoperative cisplatin-based CRT followed by esophagectomy with lymph node dissection for the locally advanced ESCC (defined by above criteria).
5. Have a performance status of 0 or 1 on the ECOG Performance Scale.
6. Exhibit at least one risk factor of tumor recurrence in the post-CRT surgical tissues:

   1. Close (≤1mm) or involved margin;
   2. Residual tumor cells in lymph nodes with extranodal invasion.
   3. ypN2 or ypN3.
7. Adequate hemogram and organ function:

   1. Absolute neutrophil count ≥1,500 /mcL; platelets ≥100,000 / mcL; hemoglobin ≥9 g/dL without transfusion or EPO dependency (within 7 days of assessment)
   2. Serum creatinine ≤1.5 X upper limit of normal or measured or calculated creatinine clearance ≥60 mL/min; serum total bilirubin ≤ 1.5 X ULN; AST and ALT ≤ 2.5 X ULN; albumin >2.5 mg/dL; international normalized ratio or prothrombin time and activated partial thromboplastin time ≤1.5 X ULN unless subject is receiving anticoagulant therapy
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female subjects of childbearing potential must be willing to use an adequate method of contraception. Contraception, for the course of the study through 120 days after the last dose of study medication.
10. Male subjects of childbearing potential must agree to use an adequate method of contraception. Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is diagnosed with adenocarcinoma of esophagus or gastroesophageal junction.
2. Has synchronously diagnosed with a squamous cell carcinoma of aero-digestive way, other than esophageal cancer.
3. Has prior malignancy, except for: (a) adequately treated basal cell or squamous cell skin cancer; (b) in-situ cervical cancer; (c) previously diagnosed malignancy which have been adequately treated and shown no evidence of recurrence for more than 5 years.
4. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
5. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
6. Has a known history of active TB (Bacillus Tuberculosis)
7. Hypersensitivity to pembrolizumab or any of its excipients.
8. Has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Hepatitis B virus positive subjects (defined as HBsAg positive and/or detectable HBV DNA).

    * Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to enrollment.
    * Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.
18. Hepatitis C virus positive subjects (defined as anti-HCV Ab positive and detectable HCV RNA).

    * Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening.
    * Participants must have completed curative anti-viral therapy at least 4 weeks prior to randomization.
19. Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and active Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.
20. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
21. Has received organ transplantation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-10-27 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-12-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hung Hsu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo JC, Huang TC, Kuo HY, Lin CC, Hsu FM, Cheng JC, Huang YL, Hsieh MS, Huang PM, Lee JM, Wu SL, Hsu CH. Adjuvant chemoradiotherapy plus pembrolizumab for locally advanced esophageal squamous cell carcinoma with high risk of recurrence following neoadjuvant chemoradiotherapy: a single-arm phase II study. Cancer Immunol Immunother. 2024 Sep 9;73(11):230. doi: 10.1007/s00262-024-03826-y. PMID 39249605
- See also: Published results — https://link.springer.com/article/10.1007/s00262-024-03826-y

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Among the 88 patients screened at National Taiwan University Hospital, Taipei City, Taiwan, between October 2018 and December 2022, 25 were finally included in the present study (protocol defined 24 evaluable patients according to statistical hypothesis and total 26 as considering for drop-out rate) .
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 25
Completed | 11
Not Completed | 14
Not completed — Lack of Efficacy | 11
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Pembrolizumab: Adjuvant cisplatin chemoradiotherapy followed by pembrolizumab
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 25
Age, Customized [Median (Full Range); unit: years]
  Median age | 62.3 [43.3 to 73.1]
Sex/Gender, Customized [Number; unit: participants]
  Male | 22
  female | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 25
Region of Enrollment [Number; unit: participants]
  Taiwan | 25

OUTCOME MEASURES:

1. Primary Outcome: 1-year Relapse-free Survival Rate
Description: From enrollment to relapse or death
Time Frame: up to 21.6 months
Population: intention-to-treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 25
months | 14.3 [9.0 to 19.5]

2. Secondary Outcome: The Median RFS
Description: from enrollment to relapse or death
Time Frame: 21.6 months
Reporting Status: Not Posted, anticipated posting 2025-05

3. Secondary Outcome: The Median Overall Survival (OS)
Description: Overall survival is from enrollment to death
Time Frame: 21.6 months
Reporting Status: Not Posted, anticipated posting 2025-05

4. Secondary Outcome: The 3-year RFS Rate
Description: Recurrence-free survival is the time from enrollment to disease recurrence or the last follow-up (censored). Recurrence will be detected by regular image study (computed scan and esophagoscopy) every 3 months during the 1st to 3rd years then every 6 months during 4th and 5th years after esophagectomy. Response Evaluation Criteria in Solid Tumors 1.1 will be used for assessment.
Time Frame: 3 years
Reporting Status: Not Posted

5. Secondary Outcome: The 3-year OS Rate.
Description: OS is the time from enrollment to death of any cause or the last follow-up (censored).
Time Frame: 3 years
Reporting Status: Not Posted

6. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability)
Description: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Time Frame: 3 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Tissue-based Biomarkers
Description: To explore the tumor tissue-based biomarkers associated with tumor recurrence.
Time Frame: 3 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Blood-based Biomarkers
Description: To explore the blood-based biomarkers associated with tumor recurrence.
Time Frame: 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: I year
Groups:
- Pembrolizumab: Pembrolizumab treatment
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 17/25
Serious Adverse Events (participants affected / at risk) | 5/25
Other Adverse Events (participants affected / at risk) | 9/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=25)
Colitis (Gastrointestinal disorders) | 1
Leucopenia (Blood and lymphatic system disorders) | 1 — during cisplatin-based chemoradiotherapy
Pancreatitis (Gastrointestinal disorders) | 1
Infection (Infections and infestations) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=25)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6
Infection (Infections and infestations) | 8
Diarrhea (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 5
Leucopenia (Blood and lymphatic system disorders) | 9 — during cisplatin-based chemoradiotherapy
anemia (Blood and lymphatic system disorders) | 5 — during cisplatin-based chemoradiotherapy
thrombocytopenia (Blood and lymphatic system disorders) | 3 — during cisplatin-based chemoradiotherapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT03322267/Prot_SAP_001.pdf